CLINICAL TRIAL: NCT06851624
Title: Six Months Follow-up of Two and Four Mini Screws Supported Hyrax for Maxillary Expansion in Non-growing Patients: A Randomized Controlled Clinical Trial
Brief Title: Six Months Follow-up of Two and Four Mini Screws Supported Hyrax in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdullah mohammed ali al-thalabi, MSc candidate, Cairo university, department of Orthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36624
Record Dates: First submitted 2025-02-12; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Transverse Maxillary Deficiency
Keywords: expansion,posterior crossbite

STUDY DESIGN:
Intervention Model Description: two experimental groups ,two screw supported and four screw supported hyrax
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one (Experimental): two mini screws supported hyrax was used
  Interventions: Device: MARPE
- Group two (Experimental): four minis crews supported hyrax was used
  Interventions: Device: MARPE

INTERVENTIONS:
Device: MARPE — treating patients with transverse maxillary deficiency using minis crews supported hybrid hyrax

SUMMARY:
six months follow-up of two and four mini-screw supported hyrax for maxillary expansion in non-growing patients: A randomized controlled clinical trial

DETAILED DESCRIPTION:
transverse malocclusion is very common in adult ,using conventional hyrax expander has many limitations and side effects such as buccal tipping, marginal bone loss, dento aloveolar expansion.

in such cases , surgically assisted rapid palatal expansion used to be the option of choice ,due to the invasiveness of the procedure and co-morbidity associated with it ,minis crews assisted rapid expansion is recently introduced to overcome the complications of both convectional and surgically assisted rapid palatal expansion

ELIGIBILITY:
Inclusion Criteria:

* adults male or female aged from 18-30 years with skeletal Maxillary constriction.
* unilateral or bilateral Dental posterior cross-bite.
* mid-palatal suture maturation (Grade C, D) according to F Angileri classification.
* good oral hygiene,

Exclusion Criteria:

* no functional crossbite due to premature contacts.
* no previous orthodontic treatment.
* no buccal crossbite.
* no craniofacial anomalies or syndromes

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Skeletal effects | 6-8 months
  To compare the amount of skeletal expansion using linear (mm) measurement extracted from cone beam computed tomography pre and post-expansion

SECONDARY OUTCOMES:
Dento-alveolar effects | 6-8 months
  To compare the amount of dento-alveolar expansion using linear (mm) measurement extracted from cone beam computed tomography pre and post-expansion
Dento-alveolar effects | 6-8 months
  To compare the amount of dento-alveolar expansion using angular(degree) measurement extracted from cone beam computed tomography pre and post-expansion

CONTACTS AND LOCATIONS:
Overall Officials: fady hussein fahim, PhD, Study Director — Associate proff; nada omar elzawahry, PhD, Study Director — lecturer; elzubair osman salih, MSc, Study Director — MSc candidates
Locations (1):
- 11,ElSaraya street ,Almanyal ,CAIRO ,EGYPT, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol